CLINICAL TRIAL: NCT06227117
Title: A Randomized, Multicenter, Open-Label Phase II Neoadjuvant Study to Evaluate the Safety and Efficacy of Disitamab Vedotin in Combination Toripalimab or Sequence Chemotherapy in Participants With HR-negative, HER2 Low-expressing Breast Cancer
Brief Title: Neoadjuvant Study of DV in Combination Toripalimab or Sequence Chemotherapy in HR-negative, HER2 Low-expressing Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC48-C024
Record Dates: First submitted 2024-01-17; First posted 2024-01-26 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-01

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; HR-negative; HER2 low-expressing
MeSH Terms: conditions — Breast Neoplasms | interventions — Carboplatin; Epirubicin; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Disitamab Vedotin + Toripalimab (Experimental): Disitamab Vedotin with Toripalimab Arm
  Interventions: Drug: Disitamab Vedotin Injection （18 weeks）; Drug: Toripalimab （18weeks）
- Disitamab Vedotin + Toripalimab+Carboplatin (Experimental): Disitamab Vedotin + Toripalimab with Carboplatin Arm
  Interventions: Drug: Disitamab Vedotin Injection （18 weeks）; Drug: Toripalimab （18weeks）; Drug: Carboplatin
- Disitamab Vedotin + Toripalimab sequential Epirubicin+ CTX+ Toripalimab (Experimental): Disitamab Vedotin + Toripalimab sequential Epirubicin+ CTX with Toripalimab Arm
  Interventions: Drug: Disitamab Vedotin Injection （12 weeks）; Drug: Sequential Epirubicin; Drug: Sequential CTX; Drug: Toripalimab （12weeks）

INTERVENTIONS:
Drug: Disitamab Vedotin Injection （18 weeks） — 2.0mg/kg, intravenous infusion，D1, every 2 weeks, Every 6 weeks is a treatment cycle. A total of 3 cycles (18 weeks) of treatment are performed.
  Other Names: DV,RC48-ADC
  Arms: Disitamab Vedotin + Toripalimab; Disitamab Vedotin + Toripalimab+Carboplatin
Drug: Toripalimab （18weeks） — 3.0 mg/kg, intravenous infusion, D1, every 2 weeks
  Other Names: JS001
  Arms: Disitamab Vedotin + Toripalimab; Disitamab Vedotin + Toripalimab+Carboplatin
Drug: Carboplatin — AUC 3 Q2W or AUC1.5 QW intravenous infusion
  Arms: Disitamab Vedotin + Toripalimab+Carboplatin
Drug: Disitamab Vedotin Injection （12 weeks） — 2.0mg/kg, intravenous infusion，D1, every 2 weeks, Every 6 weeks is a treatment cycle. A total of 2 cycles (12 weeks) of treatment are performed.
  Other Names: DV,RC48-ADC
  Arms: Disitamab Vedotin + Toripalimab sequential Epirubicin+ CTX+ Toripalimab
Drug: Sequential Epirubicin — According to body surface area, 90mg/m2, intravenous infusion, D1, every 3 weeks, A total of 12 weeks of treatment are performed.
  Other Names: Epirubicin
  Arms: Disitamab Vedotin + Toripalimab sequential Epirubicin+ CTX+ Toripalimab
Drug: Sequential CTX — According to body surface area,600mg/m2, intravenous infusion, D1, every 3 weeks, A total of 12 weeks of treatment are performed.
  Other Names: CTX, cyclophosphamide
  Arms: Disitamab Vedotin + Toripalimab sequential Epirubicin+ CTX+ Toripalimab
Drug: Toripalimab （12weeks） — 3.0 mg/kg, intravenous infusion, D1, every 2 weeks, A total of 2 cycles (12 weeks) of treatment are performed. Sequential therapy 3.0 mg/kg, intravenous infusion, D1, every 2 weeks, A total of 2 cycles (12 weeks) of treatment are performed.
  Other Names: JS001
  Arms: Disitamab Vedotin + Toripalimab sequential Epirubicin+ CTX+ Toripalimab

SUMMARY:
The purpose of this study is to evaluate the Safety and Efficacy of Neoadjuvant study of DV in combination Toripalimab i or sequence chemotherapy in HR-negative, HER2 low-expressing Breast Cancer

DETAILED DESCRIPTION:
This is an open-label, randomized, multicenter, Phase II Neoadjuvant Therapy Study designed to evaluate the Safety and Efficacy of Neoadjuvant study of DV in combination Toripalimab or sequence chemotherapy in HR-negative, HER2 low-expressing Breast Cancer The primary objectives of the study are to explore combination neoadjuvant therapy in participants with previously untreated HR-negative, HER2 low-expressing breast cancer, by assessment of tpCR and EFS.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate and sign the informed consent form;
2. Ages≥18 years;
3. Invasive breast tumour tissue with low HER2 expression confirmed by the central laboratory, defined as HER2 protein expression of IHC 1+ or IHC 2+ with no amplification by in situ hybridisation (ISH) (according to the Breast Cancer HER2 Detection Guidelines, 2019 edition) by immunohistochemistry; and specimens from the primary site of the tumour for HER2 detection (wax blocks, biopsies, or fresh tissues are acceptable) are available for HER2 detection
4. Tumour hormone receptor (HR)-negative, defined as IHC-stained invasive carcinoma with a proportion of cells positive for both ER and PgR nuclear staining of <1% according to ASCO/CAP guideline 2020;
5. Histologically confirmed invasive carcinoma of the breast according to AJCC 8th edition investigator-assessed clinical staging T1cN1-2M0, or T2-3N0-2M0
6. Subjects who tolerate and are scheduled to undergo radical breast cancer surgery and have not received any prior anti-tumour systemic therapy for breast cancer, as assessed by the research centre;
7. ECOG PS 0 or 1 point
8. At least one measurable lesion according to RECIST v1.1 criteria;
9. Cardiac function: New York Heart Association (NYHA) class <3; left ventricular ejection fraction ≥55%;
10. Bone marrow or organ function, the following criteria should be met within 7 days prior to study dosing (normal values are based on the clinical trial centre, no transfusion of blood, haematopoietic stimulating factors, albumin or blood products within 14 days prior to the test):

    1. haemoglobin ≥ 90 g/L;
    2. absolute neutrophil count (ANC) ≥ 1.5 × 109 /L;
    3. platelets ≥ 100 × 109 /L;
    4. serum total bilirubin ≤ 1.5 times the Upper Limit of Normal (ULN);
    5. Albuminous Transaminase (AST) and Albuminous Transaminase (ALT) ≤ 2.5 × ULN;
    6. International Normalised Ratio (INR) and Activated Fractional Thromboplastin Time ≤ 1.5 × ULN;
    7. Creatinine Clearance (CrCl) ≥ 60 mL/min according to the Cockcroft-Gault formula method;
11. Female subjects of childbearing potential who meet the following criteria:

    1. A serum pregnancy test (minimum sensitivity of 25 mIU/mL or equivalent units of β-human chorionic gonadotropin [β-hCG]) must be negative within 72 hours prior to the first dose of study intervention. Subjects with false-positive results and confirmed non-pregnancy will be eligible for participation in the study.
    2. Must agree to contraception for the duration of the study and for at least 6 months after the last dose of study drug .
    3. Must agree not to breastfeed or donate eggs from the time of signing the informed consent until 6 months after the last dose of study drug .
    4. If sexually active and likely to result in pregnancy, use of at least 2 acceptable contraceptive methods, at least 1 of which must be highly effective, must be continued from the time of informed consent for at least 6 months after the last dose of study drug
12. Male subjects of fertile potential who meet the following criteria:

    1. It is necessary to agree not to donate sperm from the time of signing the informed consent form until at least 4 months after the last dose of study drug.
    2. If sexual intercourse with a person of childbearing potential is likely to result in pregnancy, continuous use of at least 2 acceptable contraceptives, at least 1 of which must be highly effective, beginning at the time of informed consent and continuing until at least 4 months after the last dose of study drug. Beginning at the time of informed consent and continuing for at least 4 months after the last dose of study drug.
    3. If sex with a pregnant or breastfeeding patient, condom use must be continuous from the time of informed consent and continue until at least 4 months after the last dose of study drug.
13. Be able to understand the requirements of the trial and be willing and able to comply with the trial and follow up procedural arrangements.

Exclusion Criteria:

1. With bilateral invasive breast cancer
2. Previous history of invasive breast cancer
3. Previous carcinoma in situ of the breast with adjuvant endocrine therapy within 5 years of surgery
4. Use of investigational drugs or major surgery within 4 weeks prior to start of study drug administration
5. Live or live attenuated vaccine administered within 4 weeks prior to the start of study drug administration or planned to be administered during the study period
6. History of previous allogeneic haematopoietic stem cell transplantation or organ transplantation
7. Prior treatment with PD-(L)1, PD-L2, CTLA4 inhibitors and other antibody-coupled drugs;
8. Uncontrolled or significant cardiovascular disease, including (but not limited to): any of the following within 6 months prior to the first dose: e.g., congestive heart failure (NYHA class III or IV), myocardial infarction or cerebral infarction (except for lacunar cerebral infarction), pulmonary embolism, unstable angina, or arrhythmia requiring treatment at screening; primary cardiomyopathy (e.g., dilated cardiomyopathy, Primary cardiomyopathies (e.g., dilated cardiomyopathy, hypertrophic cardiomyopathy, arrhythmogenic right ventricular cardiomyopathy, restrictive cardiomyopathy, indeterminate cardiomyopathy); history of clinically significant prolongation of the QTc period, grade II type II AV block or grade III AV block or QTc interval (F method) >470 msec (women) or >450 msec (men); atrial fibrillation (EHRA grade ≥2b); uncontrolled hypertension that is judged by the investigator to be unsuitable; and Hypertension, judged by the investigator to be unsuitable for participation in the study;
9. History of interstitial lung disease requiring treatment or current severe lung disease including, but not limited to, active tuberculosis, interstitial lung disease;
10. Ongoing active infection that requires systemic treatment;
11. Have an active autoimmune disease requiring systemic treatment within the past 2 years (e.g., use of corticosteroids or immunosuppressive drugs, etc.), allowing for relevant replacement therapy (e.g., thyroxine, insulin, or physiological corticosteroid replacement therapy for adrenal or pituitary insufficiency)
12. A clear past or present history of a neurological or psychiatric disorder, including epilepsy or dementia
13. Ongoing grade ≥2 sensory or motor neuropathy;
14. Concomitant disease that, in the investigator's judgement, is a serious hazard to the subject's safety or interferes with the subject's ability to complete the clinical study;
15. Positive HIV test results; patients with active hepatitis B or C (HBsAg positivity accompanied by HBV DNA titres above the upper limit of normal; HCVAb positivity accompanied by HCV RNA titres above the upper limit of normal); and persistent coronavirus (COVID-19) infection.
16. Hypersensitivity reactions or delayed hypersensitivity reactions to components of Disitamab Vedotin and Toripalimab or analogues are known;
17. Known hypersensitivity or delayed hypersensitivity to epirubicin, cyclophosphamide, carboplatin preparations or components or similar drugs;
18. Other malignancy within 5 years prior to signing the informed consent (except for non-melanoma skin cancer, cervical carcinoma in situ or other tumours that have been effectively treated and are considered cured);

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-07-27 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Total pathological complete response (tpCR) rate (ypT0/Tis ypN0) | 1 month after surgery
  Defined as the proportion of participants with a pathological assessment of pCR (ypTO/Tis, ypNO) in the analyzed population;

SECONDARY OUTCOMES:
Breast pathological complete response（bpCR） | 1 month after surgery
  Defined as the proportion of participants with a pathological assessment of bpCR in the analyzed population
Objective remission rate (ORR) | Baseline to surgery
  Objective response rate.ORR assessed according to the evaluation criteria for the efficacy of solid tumors (RECIST 1.1)
Disease free survival（DFS） | Up to approximately 3 or 5 years
  From the date of surgery to the first local, regional, contralateral or distant recurrence, and death from any cause including 3- and 5-year event-free survival
Event free survival (EFS) | Up to approximately 3 or 5 years
  The time from random assignment to disease progression, including local progression before surgery; disease recurrence-local, regional, distant, ipsilateral noninvasive, or contralateral (invasive or noninvasive)-or death from any cause;
Overall survival (OS) | Date of randomization to date of death due to any cause, up to 5 years after the last subject randomized
  OS is defined as the time from the date of randomisation until the date of death due to any cause.
Adverse events | Up to approximately 2 months after surgery
  To evaluate safety including adverse event rate and adverse event grade
Change in cluster of differentiation 8 (CD8) | At baseline to surgery
  CD8 in tumor samples by biopsy at baseline and by surgery immediately after surgery would be evaluated by HE or immune staining.
Health-related quality of life - EORTC-QLQ-C30 | Up to approximately 2 years
  Change from baseline in the physical functioning subscale of the European Organisation for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) scores. Scale scores range from 0-100. For functioning and global health status/ QoL scales, higher scores indicate better functioning or global health status/QoL. For symptom scales, higher scores indicate greater symptom burden
Residual cancer burden score | 1 month after surgery
  According to the extent of the residual cancer in the primary breast cancer site (mm*mm), the residual cancer (mm*mm), cell density of residual cancer (%), proportion of carcinoma in situ (%), number of positive lymph nodes and maximum diameter of lymph node metastasis (mm), the RCB index and corresponding RCB classification can be obtained. The RCB index and the corresponding RCB grade can be obtained based on the maximum diameter of the cancer (mm).
Change in tumor-infiltrating lymphocytes (TILs) | At baseline to surgery
  Defined as infiltrating lymphocytes isolated from tumor tissue.TILs in tumor samples by biopsy right before the first neoadjuvant therapy (baseline) and by surgery immediately after surgery would be evaluated by HE or immune staining.
Change in programmed cell death protein L1 (PD-L1) | At baseline to surgery
  PD1 in tumor samples by biopsy at baseline and by surgery immediately after surgery would be evaluated by HE or immune staining.

CONTACTS AND LOCATIONS:
Overall Officials: Changling Li, Study Director — RemeGen Co., Ltd.
Locations (5):
- China (5):
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No